CLINICAL TRIAL: NCT03779880
Title: Examining Parkinson's Disease-Related Retirement: Results of Turkey
Status: Completed | Type: Observational
Sponsor: Istanbul Kültür University (Other)
Collaborators: Marmara University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Gamze Ertürk, Research assistant, Istanbul Kültür University
Other Study IDs: 132
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease, Early Retirement,
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Although Parkinson Disease's (PD) is usually associated with an older patient population, 5% of patients are diagnosed at age 50 and 30% before 65 years of age. This shows that many patients with PD have diagnosed during the active study and have long periods of normal retirement. After the diagnosis of Parkinson's patients, the duration of leaving of employment vary between 0 and 25 years. It was found that patients' full-time working capacity decreased by up to 80% and they quitted earlier than the general population. The disability associated with PD is thought to be a factor in this situation. Nevertheless, the reasons for early retirement are not fully known and more information is needed on the specific problems of PD in order for patients to continue their career. The aim of our study is to examine the impact of Parkinson's disease on retirement and to contribute to Turkey's data. Patients with PD admitted to the Parkinson's disease outpatient clinic, which is the biggest clinic of Turkey about neurology, are included in the study. It is planned to meet with 75 patients on 31/12/2018 and to reach the end of the data collection phase.

ELIGIBILITY:
Inclusion Criteria:

* To be between 30-85 aged
* Parkinson Disease diagnosis according to the United Kingdom Brain Bank criteria
* To be treated with antiparkinson

Exclusion Criteria:

* Dementia
* Severe cognitive impairment
* Not willing to participate in the study

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were chosen from among retired Parkinson's patients who met the inclusion criteria and are applied Istanbul Cerrahpaşa University, has largest movement disorders unit of Turkey, between May and December 2018.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-03-28 (Actual)

PRIMARY OUTCOMES:
Qualitative interview | The researcher interviewed for about half an hour at once time with each participant.
  The researcher conducted interviews to find out about things that could not be directly observed. Interviews have been done face to face and used to collect personal experiences about Parkinson Disease and work life.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Ertürk, GRAD ASST, Study Chair — Istanbul Kültür University; Semra Oğuz, ASST PROF, Study Director — Marmara University
Locations (1):
- Istanbul Cerrahpaşa University, Istanbul, Turkey (Türkiye)